CLINICAL TRIAL: NCT03475277
Title: Mapping the Influence of Drugs of Abuse on Risk and Reward Circuits
Brief Title: Stanford Regulating Circuits of the Brain Study- Ketamine
Acronym: RBRAIN-KET
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Leanne Williams, Professor of Psychiatry and Behavioral Sciences, Stanford University
Other Study IDs: 41173; 1P50DA042012-01A1 (NIH)
Record Dates: First submitted 2018-03-01; First posted 2018-03-23 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Healthy
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Volunteers: Participants will receive an IV infusion of ketamine (~.05mg/kg and 0.5mg/kg) or placebo.
  Ketamine is an FDA-approved dissociative anesthetic. The study doses are in the subanesthetic range. During the infusion, an ACLS-certified psychiatrist or anesthesiologist will provide continuous monitoring.
  Afterwards, patients will be monitored on-site by an ACLS-certified MD or highly skilled research nursing staff, and an on-call emergency response team for 4 hours (ketamine's half-life is 15 min; 4 hrs= 16 half-lives).
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Acute administration
  Other Names: "special k"

SUMMARY:
This study is a biomarker study designed to characterize how ketamine impacts the reward circuits of the human brain.

DETAILED DESCRIPTION:
The investigators will assess the effect of acute ketamine modulation on the functioning of reward-related human brain circuits. Reward-related brain circuits will be assessed using functional magnetic resonance imaging.

Participants will include volunteers who report more than two prior uses of ketamine (also known as "Special K"), when they were 18 years or older.

The investigators will recruit individuals who have previously tried ketamine rather than those who are ketamine-naïve.

Participants will receive an IV infusion of ketamine (~.05mg/kg and 0.5mg/kg) or placebo (saline). Following established procedures, these three sessions will be randomized in a blinded protocol in order to limit expectancy effects.

Throughout each session, participants will be monitored. Functional imaging will commence after the drug has reached peak levels, following previously established time courses for ketamine infusion. Participants will also be monitored after the functional imaging session. Secondary effects of ketamine on behavior and self-reported experience will be assessed.

In the assessment of the acute effects of ketamine, the investigators will take into account the cumulative effects of prior drug exposure.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-55 years
* At least 2 prior uses of ketamine when aged 18+
* BMI within healthy range (18-30)
* Ability to speak, read, or understand English

Exclusion Criteria:

* Current active suicide ideation or history of suicide attempts
* Current mood, anxiety, eating, psychotic, or substance use disorder
* Lifetime psychotic or bipolar disorder
* Schizophrenia in a first degree relative
* Current use of psychotropic medication
* Prior adverse ketamine response
* Allergy or hypersensitivity to ketamine
* Use of ketamine in past 7 days
* Cannabis use in the past 7 days, illicit recreational drug use in the 48 hours prior to sessions, and/or alcohol use in the 24 hours prior to sessions
* Concurrent use of any medications that might increase the risk of participation (e.g., drug interactions)
* History of epilepsy, convulsions, seizures, LOC >10 min
* Renal/hepatic impairment
* Hypertension (Stage 1 defined as systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg on 2 of 3 measurements at least 15 min apart at initial screening; systolic blood pressure >155 mmHg or diastolic blood pressure >99 mmHg on 2 of 3 measurements at least 15 min apart during infusion visits)
* Heart rate <50 bpm or >150 bpm at initial screening
* Chronic congestive heart failure, tachyarrhythmias, myocardial ischemia assessed via EKG at initial screening
* EKG QTcF intervals >430 ms for men and >470 ms for women
* Direct physical access to or routine handling of addicting drugs in the regular course of work duties
* MRI contraindication
* Pregnant or nursing females

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Healthy volunteers with prior exposure to ketamine
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Circuit activation as assessed by functional magnetic resonance imaging | Up to 2 weeks after infusion of ketamine or placebo
  During functional magnetic resonance imaging the reward and negative affect circuits will be engaged by reward and related emotional tasks, and circuit activation will be quantified by blood flow in regions of interest and the extent of functional connectivity between them

SECONDARY OUTCOMES:
Behavioral responses on the WebNeuro computerized test battery assessing cognitive capacity | Up to 5 hours after infusion of ketamine or placebo
  Accuracy data are quantified as number of errors and lower values indicate better performance
Self-reported responses as assessed by the 21-item Depression, Anxiety and Stress Scale (DASS) | Up to 5 hours after infusion of ketamine or placebo
  Responses are quantified on a 4-point scale and summed for total DASS score and for each Depression, Anxiety and Subscale score. Higher scores indicate more severe symptoms of depression, anxiety and stress
Level of subjectively experienced intoxication, dissociation, and mood and feelings as assessed by rating scale. | Up to 5 hours after infusion of ketamine or placebo
  Responses will be quantified in intervals of 10 on a visual analogue of 1 to 100
Self-reported responses as assessed by the 29-item Rotter's Locus of Control (RLoC) | Up to 5 hours after infusion of ketamine or placebo
  Responses are quantified as a summed score from 0 to 23 and determine the degree to which a person perceives an outcome as being contingent on their own actions or those of external forces. Higher scores indicate greater levels of external locus of control.
Self-reported responses as assessed by the 15-item Mini Brief Risk-Resilience Index for Screening (BRISC). | Up to 5 hours after infusion of ketamine or placebo
  Responses are quantified on a 5-point Likert scale and is a measure of emotional self-regulation. Scores measure three core domains: negativity bias, emotional resilience, and social skills. Higher scores indicate higher functioning and better coping.
Self-reported responses as assessed by the 14-item Snaith-Hamilton Please Scale (SHAPS). | Up to 5 hours after infusion of ketamine or placebo
  Responses are quantified on a 4-point scale and measures anhedonia, the inability to experience pleasure. Scores measure domains of social interaction, food and drink, sensory experience, and interest/pastimes. An "abnormal" score is defined as 3 or more.
Self-reported responses as assessed by the 24-item Dimensional Apathy Scale (DAS). | Up to 5 hours after infusion of ketamine or placebo
  Responses are quantified on a 4-point scale and measure demotivation in three domains: executive apathy, emotional apathy, and initiation apathy. Higher scores indicate higher apathy level.
Self-reported responses as assessed by the 18-item Motivation and Pleasure Scale Self-Report (MAP-SR). | Up to 5 hours after infusion of ketamine or placebo
  Responses are quantified on a 5-point Likert scale and assesses an individual's motivation and pleasure. Higher scores indicate higher levels of motivation and pleasure.
Self-reported responses as assessed by the 17-item Dimensional Anhedonia Rating Scale (DARS). | Up to 5 hours after infusion of ketamine or placebo
  Responses are summed on a 5-point scale. Scores assess interest, motivation, effort, and consummatory pleasure across four domains: hobbies, food/drink, social activities, and sensory experiences. Lower scores represent a higher level of anhedonia.
Self-reported responses as assessed by the 94-item 5-Dimensional Altered States of Consciousness Rating Scale (DASC). | Up to 5 hours after infusion of ketamine or placebo
  Responses are recorded on a sliding scale with one side reading 'No, not more than usually' and the opposite reading 'Yes, much more than usually'. More agreeance to the statements represents that the individual is experiencing higher levels of altered states of consciousness.
Self-reported responses as assessed by the 23-item Clinician Administered Dissociative States Scale (CADSS). | Up to 5 hours after infusion of ketamine or placebo
  Responses are summed on a 5-point scale in rating one's agreeance to the dissociative statements as 'not at all' to 'extreme'. Scores assess individual's dissociative state. A higher score represents more dissociation.
Self-reported responses as assessed by a clinician on the 18-item Brief Psychiatric Rating Scale (BPRS). | Up to 5 hours after infusion of ketamine or placebo
  Responses are summed on a 7-point scale in rating one's severity to the statements as 'not assessed' to 'extremely severe'. Scores assess psychiatric symptoms like anxiety, depression, and psychoses. A higher score means the individual is presenting more extreme symptoms.
Steroid hormone assay via saliva collection | Up to 5 hours after infusion of ketamine or placebo
  At 5 different time points throughout infusion visits the participant chews on a cotton swab for 30 seconds to collect saliva. A steroid hormone assay is conducted to collect data on cortisol, testosterone, progesterone, and estradiol levels.

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Williams, PhD, Principal Investigator — Study PI
Locations (1):
- Stanford Psychiatry, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hack LM, Zhang X, Heifets BD, Suppes T, van Roessel PJ, Yesavage JA, Gray NJ, Hilton R, Bertrand C, Rodriguez CI, Deisseroth K, Knutson B, Williams LM. Ketamine's acute effects on negative brain states are mediated through distinct altered states of consciousness in humans. Nat Commun. 2023 Oct 19;14(1):6631. doi: 10.1038/s41467-023-42141-5. PMID 37857620
- See also: Link to results reference — https://www.nature.com/articles/s41467-023-42141-5